CLINICAL TRIAL: NCT03283020
Title: Opioid-Induced Swallowing Dysfunction - The Impact of Bolus Volume: a Randomized, Double-Blind Study in Healthy Volunteers
Brief Title: Opioid-Induced Swallowing Dysfunction - The Impact of Bolus Volume
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Johanna Savilampi, MD, PhD, Region Örebro County
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JS006
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Pharyngeal Dysfunction; Pharyngeal Swallowing
Keywords: Remifentanil; Methylnaltrexone; Pharyngeal dysfunction; Anesthetic sedation
MeSH Terms: interventions — methylnaltrexone; Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RemifentanilMNTX (Active Comparator): Volunteers are given an intravenous infusion with remifentanil, with an effect-site target concentration of 3 ng/ml via a target-controlled infusion (TCI) pump. After a series of swallowing tests an intravenous injection of methylnaltrexone of 0,3 mg/kg is given.
  Interventions: Drug: RemifentanilMNTX
- PlaceboMNTX (Active Comparator): Volunteers are given an intravenous infusion with saline 0,9%. After a series of swallowing tests an intravenous injection of methylnaltrexone of 0,3 mg/kg is given.
  Interventions: Drug: PlaceboMNTX

INTERVENTIONS:
Drug: RemifentanilMNTX — Remifentanil infusion TCI 3 ng/ml, Methylnaltrexone injection 0.3 mg/kg
  Other Names: Methylnaltrexone; Remifentanil; Relistor; Ultiva
  Arms: RemifentanilMNTX
Drug: PlaceboMNTX — Placebo (NaCl 0.9%) TCI infusion, Methylnaltrexone injection 0.3 mg/kg
  Other Names: Sodium Chloride 0.9%; Methylnaltrexone; Relistor
  Arms: PlaceboMNTX

SUMMARY:
The purpose of the study is to evaluate the impact of different bolus volumes and viscosity on remifentanil-induced swallowing dysfunction in healthy volunteers.Hence, whether swallowing tasks can be done safer during sedation by altering bolus volumes and viscosities will be revealed. Furthermore, the study will clarify underlying mechanisms (central vs. peripheral effects) of remifentanil-induced swallowing dysfunction. If methylnaltrexone reverses the remifentanil-induced effects on swallowing, this would suggest a dominant peripherally mediated mechanism.

DETAILED DESCRIPTION:
Monitored anesthesia care (MAC) is commonly applied in modern perioperative care and means that minor surgical procedures are accomplished in awake patients using local anesthesia and light sedation. MAC has many advantages compared to general anesthesia; the recovery time after anesthesia is shorter and risk for postoperative nausea is lower to mention some. However, the patient is spontaneously breathing and the airway is not protected by an endotracheal tube which potentially increases risk of pulmonary aspiration. Pulmonary aspiration, that is inhalation of stomach and/or pharyngeal contents into the lungs, is a severe anesthesia-related complication and can in worst case lead to pneumonia and even death. Intact swallowing function is crucial in avoiding aspiration and how sedatives and analgesic agents used during MAC influence swallowing function is not fully understood.

Pharyngeal function during bolus swallowing is measured by combined high resolution impedance manometry (HRIM). The HRIM catheter is inserted through the nose in such a way that sensors straddle the entire pharynx and esophagus with the distal catheter tip in the stomach. Dynamic pressure changes and flow can be detected during swallowing and data registered by HRIM are analysed using purpose-designed software, AIM analysis (automated impedance manometry analysis). AIM analysis derives pressure flow variables which describe different physiological events like bolus timing and bolus distension in the pharynx and the esophagus during swallowing. A Swallow Risk Index value, quantifying risk of deglutitive aspiration, can also be defined.

The aim of the study is to evaluate impact of different bolus volumes on remifentanil-induced swallowing dysfunction in healthy volunteers. The study will clarify underlying mechanisms (central vs. peripheral effects) of remifentanil-induced swallowing dysfunction. Furthermore, whether swallowing tasks can be done safer during sedation by altering bolus volumes will be revealed. In addition to bolus volume, different bolus viscosities will be tested. It is shown that higher bolus viscosity diminishes misdirected swallows in dysphagic patients and higher bolus viscosity may possibly counteracts the swallowing dysfunction induced by remifentanil. Moreover, if MNTX reverses the remifentanil-induced effects on swallowing, then this would suggest a dominant peripherally mediated mechanism. Our aim is also to evaluate impact of remifentanil exposure on esophageal motility and impact of methylnaltrexone alone on swallowing function.

20 healthy volunteers will be studied on two different occasions approximately one week apart. In a randomized order volunteers will receive intravenous infusion of remifentanil and an intravenous injection of MNTX on one occasion, and placebo (normal saline) infusion and an intravenous injection of MNTX on the other occasion. Blood samples are obtained for plasma concentration determination of the study drug and sedation levels are assessed during study drug exposure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 - ≤ 40 year old healthy volunteers from both sexes.
2. Have signed and dated Informed Consent.
3. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Anamnesis of pharyngoesophageal dysfunction.
2. Known or history of gastrointestinal, severe cardiac, pulmonary or neurological disease
3. Ongoing medication that may affect upper gastrointestinal tract, larynx or lower airway.
4. Allergies to or history of reaction to remifentanil, fentanyl analogues or dexmedetomidine.
5. Pregnancy or breast feeding
6. BMI > 30
7. Smoking
8. Previous participation in a medicinal clinical trial during the last year where an opioid has been used or have during the last 30 days participated in any other medicinal clinical trial or in a trial where follow-up is not completed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Pressure Flow pharyngeal variables, 10 ml vs 20 ml bolus | Up to 60 minutes
  Difference in pharyngeal pressure flow variables during remifentanil exposure between bolus volumes of 10 ml and 20 ml compared to placebo.

SECONDARY OUTCOMES:
Pressure Flow pharyngeal variables, liquid vs semisolid bolus | Up to 60 minutes
  Difference in pharyngeal pressure flow variables during remifentanil exposure between liquid and semisolid boluses compared to placebo
Pressure Flow pharyngeal variables, remifentanil before vs after methylnaltrexone | Up to 60 minutes
  Difference in pharyngeal pressure flow variables during remifentanil exposure before and after methylnaltrexone administration compared to placebo.
Pressure Flow pharyngeal variables, placebo before vs after methylnaltrexone | Up to 60 minutes
  Difference in pharyngeal pressure flow variables during placebo infusion before and after methylnaltrexone administration.
Pressure Flow esophageal motility variables, 10 ml vs 20 ml bolus | Up to 60 minutes
  Difference in variables of esophageal motility between different bolus volumes during remifentanil exposure compared to placebo.
Pressure Flow esophageal motility variables, liquid vs semisolid bolus | Up to 60 minutes
  Difference in variables of esophageal motility between liquid and semisolid boluses during remifentanil exposure compared to placebo.
Pressure Flow esophageal motility variables, remifentanil before vs after methylnaltrexone | Up to 60 minutes
  Difference in variables of esophageal motility during remifentanil exposure before and after methylnaltrexone administration compared to placebo.
Pressure Flow esophageal motility variables, placebo before vs after methylnaltrexone | Up to 60 minutes
  Difference in variables of esophageal motility during placebo infusion before and after methylnaltrexone administration.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Savilampi, MD, PhD, Principal Investigator — University hospital in Örebro
Locations (1):
- Department of Anaesthesiology and Intensive Care, Örebro University Hospital, Örebro, Sweden